CLINICAL TRIAL: NCT04127487
Title: Quantification of NLRP3 (rs4612666) and CARD8 Gene (rs2043211) in Subgingival Plaque and Blood Samples of Generalized Chronic Periodontitis Subjects With and Without Coronary Heart Disease
Brief Title: Quantification of NLRP3 (rs4612666) and CARD8 Gene (rs2043211) in Generalized Chronic Periodontitis Subjects
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Meenakshi Ammal Dental College and Hospital (Other)
Responsible Party: Principal Investigator, Dr.Jaideep Mahendra, Professor and PhD guide, Meenakshi Ammal Dental College and Hospital
Other Study IDs: MADC/IRB-XXV/2018/391
Record Dates: First submitted 2019-10-14; First posted 2019-10-15 (Actual); Last update posted 2019-12-03 (Actual); Status verified 2019-12

CONDITIONS: Periodontal Diseases; Coronary Artery Disease
Keywords: NLRP3 (rs4612666), CARD8 (rs20432111)
MeSH Terms: conditions — Periodontal Diseases; Coronary Artery Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Periodontitis group: 35 Generalized chronic periodontitis subjects without coronary heart diseases
- periodontitis with CAD group: 35 Generalized chronic periodontitis subjects diagnosed with Coronary heart disease

SUMMARY:
Quantification of NLRP3 (rs4612666) and CARD8 (rs20432111) will be analysed in the subgingival plaque and blood samples of generalized chronic periodontitis with and without coronary heart disease. The demographic and the periodontal parameters were assessed and correlated with the quantification of NLRP3 (rs4612666) and CARD8 (rs2043211) was analysed with RT-PCR

DETAILED DESCRIPTION:
The study is done in order to assess the demographic variables such as age, height, weight and socio-economic status, BMI, personal habits, waist-hip ratio, lipid profile, use of medications, and family history of coronary artery disease in generalised chronic periodontitis subjects with and without coronary artery disease. To assess and compare the periodontal status of generalised chronic periodontitis subjects with and without coronary artery disease. To determine the expression of NLRP3 (rs4612666) and CARD8 gene (rs2043211) polymorphisms in subgingival tissue samples of generalised chronic gingivitis periodontitis subjects with and without coronary artery disease. To correlate the demographic variables and periodontal parameters and the expression of NLRP3 (rs4612666) and CARD8 (rs2043211) gene polymorphisms in generalised chronic periodontitis patients with coronary artery disease and compare them with systemically healthy chronic periodontitis patients

ELIGIBILITY:
Inclusion Criteria:

* Patients willing to participate in the study
* Patients within the age group of 30-65 years ( male )
* Patients should have ≥ 20 remaining natural teeth
* No history of long term antibiotic use in the past 6 months
* For group I generalized chronic periodontitis patients with coronary heart disease
* For group II generalized chronic periodontitis patients without coronary heart disease

Exclusion criteria:

* Patients with systemic conditions such as type I, and type II diabetes mellitus, respiratory diseases, renal disease, liver disease, rheumatoid arthritis, allergy, advanced malignancies and hiv infection will be excluded from the present investigation.
* Patients on drugs such as corticosteroids, antibiotics within 3 months of investigation will be excluded.
* Current smokers, individuals who quit smoking less than 6 months ago.
* Patients who had undergone periodontal therapy within the previous 6 months

Ages: 30 Years to 65 Years | Sex: Male
Age Groups: Adult, Older Adult
Gender Based: Yes — Only male patients in the age group of 30-65 years were included. Females were excluded due to hormonal changes or pregnancy that may alter the oral flora
Study Population: All male patients within the age group of 30-65 years. The subjects were from south indian population
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2019-10-01 (Actual); Primary Completion 2020-11-01 (Estimated); Study Completion 2020-12-01 (Estimated)

PRIMARY OUTCOMES:
Expression of NLRP3 (rs4612666) and CARD8 (rs20432111) gene | 12 months
  Expression of NLRP3 (rs4612666) and CARD8 (rs20432111) gene using RT-PCR

SECONDARY OUTCOMES:
Quantification of NLRP3 (rs4612666) and CARD8 (rs20432111) gene | 12 months
  Quantification of NLRP3 (rs4612666) and CARD8 (rs20432111) gene using RT-PCR

CONTACTS AND LOCATIONS:
Overall Officials: Jaideep Mahendra, MDS, PhD, Study Director — Meenakshi Ammal Dental College
Locations (1):
- Jaideep Mahendra, Chennai, Tamil Nadu, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Isaza-Guzman DM, Hernandez-Viana M, Bonilla-Leon DM, Hurtado-Cadavid MC, Tobon-Arroyave SI. Determination of NLRP3 (rs4612666) and IL-1B (rs1143634) genetic polymorphisms in periodontally diseased and healthy subjects. Arch Oral Biol. 2016 May;65:44-51. doi: 10.1016/j.archoralbio.2016.01.013. Epub 2016 Jan 27. PMID 26854620